CLINICAL TRIAL: NCT01823432
Title: Genetic Risks for Bicuspid Aortic Valve Disease
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Siddharth Prakash, Assistant Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-11-0185
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Bicuspid Aortic Valve; Unicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; unicuspid aortic valve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Genomic DNA from whole blood Genomic DNA from saliva Aortic valve tissue preserved in RNALater
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAV Cohort: Patients with bicuspid or unicuspid aortic valves, regardless of surgical status.

SUMMARY:
Bicuspid Aortic Valve (BAV) is the most common congenital heart malformation in adults, but very little is known about the genetic causes or risk factors for adverse outcomes. Currently, it is estimated that most cases of aortic stenosis in patients less than 65 years old are caused by BAVs. BAV patients are also at high risk to develop aneurysms of the ascending aorta, which may lead to aortic dissections. Dr. Prakash and his colleagues plan to use individual genetic information to identify persons with BAV who are at high risk for complications and to customize therapies.

DETAILED DESCRIPTION:
To be included in the study, patients must have a bicuspid or unicuspid aortic valve, documented by clinical history or imaging studies. If the aortic valve was replaced surgically, they may still be eligible. Participants will be asked to donate a single tube of blood and fill out a questionnaire. Patients will also be followed up by telephone or email about once a year to determine if they experience any medical complications related to Bicuspid Aortic Valve (BAV), such as aortic aneurysms, aortic dissections or valve disease. Patients may not be included if they are less than 18 years old at the time of recruitment or have a recognized genetic syndrome or genetic mutation such as Marfan or Ehlers-Danlos syndrome.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of bicuspid or unicuspid aortic valve

Exclusion Criteria:

* Less than 18 years of age
* Recognized syndrome or identified genetic mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults at least 18 years old with unicuspid or bicuspid aortic valves
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Thoracic aortic aneurysms and dissections | 10 years
  Development of new aneurysms and/or dissections of the thoracic aorta
Aortic valve replacement surgery | 10 years

SECONDARY OUTCOMES:
Aortic enlargement | 10 years
  Dilation of thoracic aorta, new or progressive

OTHER OUTCOMES:
Aortic valve degeneration | 10 years
  Increase in valve degeneration score by at least 1 unit

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Prakash, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DiGregorio H, Mansoorshahi S, Carlisle SG, Tovar Pensa C, Watts A, McNeely C, Sabate-Rotes A, Yetman A, Michelena HI, De Backer JFA, Mosquera LM, Bissell MM, Andreassi MG, Foffa I, Hui DS, Caffarelli A, Kim YY, Citro R, De Marco M, Tretter JT, McBride KL, Body SC, Milewicz DM, Prakash SK; EBAV Investigators. Contribution of rare chromosome 22q11.2 copy number variants to non-syndromic bicuspid aortic valve. Heart. 2025 Feb 12;111(5):221-229. doi: 10.1136/heartjnl-2024-324669. PMID 39658198
- See also: John Ritter Research Program in Aortic and Vascular Disease — http://www.johnritterresearchprogram.org/